CLINICAL TRIAL: NCT00848718
Title: A Phase I Dose Escalation Study of MK-2206 in Combination With Standard Doses of Selected Chemotherapies or Targeted Agents in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Phase I Study of MK-2206 in Combination With Standard Chemotherapy in Participants With Locally Advanced or Metastatic Solid Tumors (MK-2206-003)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2206-003; 2009_547; MK-2206-003 (Other: Merck)
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Results first posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Locally Advanced, Metastatic Solid Tumors
Keywords: Tumors, cancer
MeSH Terms: conditions — Neoplasms | interventions — MK 2206; Docetaxel; Erlotinib Hydrochloride; Carboplatin; Paclitaxel; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MK-2206 + carboplatin + paclitaxel (Experimental): MK-2206 combined with carboplatin and paclitaxel
  Interventions: Drug: MK-2206; Drug: carboplatin; Drug: paclitaxel
- MK-2206 + docetaxel (Experimental): MK-2206 combined with docetaxel plus pretreatment with a corticosteroid
  Interventions: Drug: MK-2206; Drug: docetaxel; Drug: corticosteroid
- MK-2206 + erlotinib (Experimental): MK-2206 combined with erlotinib
  Interventions: Drug: MK-2206; Drug: erlotinib

INTERVENTIONS:
Drug: MK-2206 — MK-2206 given by mouth (PO) on Days 1, 3, 5, and 7 of each 21-day cycle (30 mg, 45 mg, or 60 mg) OR MK-2206 PO on Day 1 of each 21-day cycle (60 mg, 90 mg, 135 mg, 200 mg , or 250 mg)
Drug: docetaxel — Administered as an IV infusion on Day 1 of each 21-day cycle
  Other Names: Taxotere®
  Arms: MK-2206 + docetaxel
Drug: erlotinib — Administered daily (QD) PO in each 21-day cycle
  Other Names: Tarceva®
  Arms: MK-2206 + erlotinib
Drug: carboplatin — Administered as an intravenous (IV) infusion on Day 1 of every 21-day cycle
  Other Names: Paraplatin®
  Arms: MK-2206 + carboplatin + paclitaxel
Drug: paclitaxel — Administered as an intravenous (IV) infusion on Day 1 of every 21-day cycle
  Other Names: Taxol®
  Arms: MK-2206 + carboplatin + paclitaxel
Drug: corticosteroid — Administered PO twice a day (BID) on Days 1-3 of each 21-day cycle
  Arms: MK-2206 + docetaxel

SUMMARY:
The purpose of this study is to compare the safety and tolerability of several dose levels of MK-2206 in combination with chemotherapy and targeted therapy agents in participants with locally advanced or metastatic solid tumors.

The primary hypotheses are that administration of MK-2206 in combination with either carboplatin + paclitaxel, docetaxel, or erlotinib in participants with locally advanced or metastatic solid tumors will have acceptable tolerability, a dose limiting toxicity (DLT) rate of ≤30%, plasma exposure and pharmacodynamics that exceed target thresholds, and allow for definition of a maximum tolerated dose (MTD) in each of the 3 combinations.

ELIGIBILITY:
Inclusion Criteria :

* Participants must have locally advanced or metastatic solid tumors.
* Participant is male or female greater than or equal to 18 years of age.
* Participant must have a performance status less than or equal to 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
* Female participants of childbearing potential has a negative serum or urine pregnancy test within 72 hours prior to receiving the first dose of study medication.
* Participants in the MK-2206 + carboplatin/paclitaxel and MK-2206 + docetaxel treatment arms will be limited to no more than 3 prior cytotoxic therapies for metastatic or recurrent diseases.
* Participant is able to swallow capsules and has no surgical or anatomical condition that will prevent the Participant from swallowing.

Exclusion Criteria:

* Participant has had chemotherapy, radiotherapy or biological therapy within 4 weeks.
* Participants must be least 4 weeks post-surgery and do not expect major surgery in the study duration.
* Participant is currently participating or has participated in a study with an investigational compound or device within 30 days.
* Participant has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Participant with a primary central nervous system tumor.
* Participant has known hypersensitivity to the components of study drug.
* Participant has a history or current evidence of heart disease.
* Participant has evidence of clinically significant bradycardia (slow heart rate).
* Participant has uncontrolled high blood pressure.
* Participant at significant risk for hypokalemia (low potassium levels).
* Participant is a known diabetic
* Participant has known psychiatric or substance abuse disorders.
* Participant is a user of illicit drugs.
* Participant is pregnant or breastfeeding.
* Participant is Human Immunodeficiency Virus (HIV) positive.
* Participant has known history of Hepatitis B or C or active Hepatitis A.
* Participant has symptomatic ascites or pleural effusion.
* Participant is receiving treatment with oral corticosteroids.
* Participant is using a potent cytochrome P(450) 3A4 (CYP3A4) inhibitor or inducer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2009-03-17 (Actual); Primary Completion 2011-05-19 (Actual); Study Completion 2012-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Molife LR, Yan L, Vitfell-Rasmussen J, Zernhelt AM, Sullivan DM, Cassier PA, Chen E, Biondo A, Tetteh E, Siu LL, Patnaik A, Papadopoulos KP, de Bono JS, Tolcher AW, Minton S. Phase 1 trial of the oral AKT inhibitor MK-2206 plus carboplatin/paclitaxel, docetaxel, or erlotinib in patients with advanced solid tumors. J Hematol Oncol. 2014 Jan 3;7:1. doi: 10.1186/1756-8722-7-1. PMID 24387695

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 77 participants were allocated to one of 3 treatment combinations with MK-2206 according to clinical presentation but 5 participants were not treated due to disease progression before initiation of treatment.
Groups:
- MK-2206 45 mg QOD+Carboplatin+Paclitaxel: Participants received MK-2206 45 mg administered PO on Days 1, 3, 5, and 7 in combination with carboplatin AUC 6 and paclitaxel 200 mg/m^2 administered IV on Day 1 of each 21-day cycle.
- MK-2206 60 mg QOD+Carboplatin+Paclitaxel: Participants received MK-2206 60 mg administered PO on Days 1, 3, 5, and 7 in combination with carboplatin AUC 6 and paclitaxel 200 mg/m^2 administered IV on Day 1 of each 21-day cycle.
- MK-2206 90 mg Q3W+Carboplatin+Paclitaxel: Participants received MK-2206 90 mg administered PO in combination with carboplatin AUC 6 and paclitaxel 200 mg/m^2 administered IV on Day 1 of each 21-day cycle.
- MK-2206 135 mg Q3W+Carboplatin+Paclitaxel: Participants received MK-2206 135 mg administered PO in combination with carboplatin AUC 6 and paclitaxel 200 mg/m^2 administered IV on Day 1 of each 21-day cycle.
- MK-2206 200 mg Q3W+Carboplatin+Paclitaxel: Participants received MK-2206 200 mg administered PO in combination with carboplatin AUC 6 and paclitaxel 200 mg/m^2 administered IV on Day 1 of each 21-day cycle.
- MK-2206 45 mg QOD+Docetaxel 75 mg/m^2: Participants received MK-2206 45 mg administered PO on Days 1, 3, 5, and 7 in combination with Docetaxel 75 mg/m^2 administered IV on Day 1 of each 21-day cycle. Participants also received an oral corticosteroid PO daily.
- MK-2206 90 mg Q3W+Docetaxel 60 mg/m^2: Participants received MK-2206 90 mg administered PO on Day 1 in combination with Docetaxel 60 mg/m^2 administered IV on Day 1 of each 21-day cycle. Participants also received an oral corticosteroid PO daily.
- MK-2206 135 mg Q3W+Docetaxel 60 mg/m^2: Participants received MK-2206 135 mg administered PO on Day 1 in combination with Docetaxel 60 mg/m^2 administered IV on Day 1 of each 21-day cycle. Participants also received an oral corticosteroid PO daily.
- MK-2206 200 mg Q3W+Docetaxel 60 mg/m^2: Participants received MK-2206 200 mg administered PO on Day 1 in combination with Docetaxel 60 mg/m^2 administered IV on Day 1 of each 21-day cycle. Participants also received an oral corticosteroid PO daily.
- MK-2206 45 mg QOD+Erlotinib 100 mg: Participants received MK-2206 45 mg administered PO every other day (Days 1, 3, 5, 7, 9, 11, 13, 15, 17, 19 and 21) in combination with Erlotinib 100 mg administered PO once every day of each 21-day cycle.
- MK-2206 45 mg QOD+Erlotinib 150 mg: Participants received MK-2206 45 mg administered PO every other day (Days 1, 3, 5, 7, 9, 11, 13, 15, 17, 19 and 21) in combination with Erlotinib 150 mg administered PO once every day of each 21-day cycle.
- MK-2206 135 mg QW+Erlotinib 100 mg: Participants received MK-2206 135 mg administered PO on Days 1, 8 and 15 in combination with Erlotinib 100 mg administered PO once every day of each 21-day cycle.
- MK-2206 135 mg QW+Erlotinib 150 mg: Participants received MK-2206 135 mg administered PO on Days 1, 8 and 15 in combination with Erlotinib 150 mg administered PO once every day of each 21-day cycle.
Period: Overall Study
Arm/Group | MK-2206 45 mg QOD+Carboplatin+Paclitaxel | MK-2206 60 mg QOD+Carboplatin+Paclitaxel | MK-2206 90 mg Q3W+Carboplatin+Paclitaxel | MK-2206 135 mg Q3W+Carboplatin+Paclitaxel | MK-2206 200 mg Q3W+Carboplatin+Paclitaxel | MK-2206 45 mg QOD+Docetaxel 75 mg/m^2 | MK-2206 90 mg Q3W+Docetaxel 60 mg/m^2 | MK-2206 135 mg Q3W+Docetaxel 60 mg/m^2 | MK-2206 200 mg Q3W+Docetaxel 60 mg/m^2 | MK-2206 45 mg QOD+Erlotinib 100 mg | MK-2206 45 mg QOD+Erlotinib 150 mg | MK-2206 135 mg QW+Erlotinib 100 mg | MK-2206 135 mg QW+Erlotinib 150 mg
Started | 7 | 9 | 6 | 5 | 6 | 5 | 3 | 5 | 4 | 9 | 4 | 6 | 8
Treated | 6 (1 participant was allocated but did not receive treatment due to progression of disease) | 9 | 5 (1 participant was allocated but did not receive treatment due to progression of disease) | 5 | 6 | 5 | 3 | 4 (1 participant was allocated but did not receive treatment due to progression of disease) | 4 | 9 | 4 | 6 | 6 (2 participants were allocated but did not receive treatment due to progression of disease)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 9 | 6 | 5 | 6 | 5 | 3 | 5 | 4 | 9 | 4 | 6 | 8
Not completed — Adverse Event | 2 | 2 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 1
Not completed — Progressive disease before treatment | 1 | 5 | 1 | 3 | 4 | 4 | 2 | 1 | 2 | 7 | 3 | 6 | 2
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Progressive disease during treatment | 3 | 0 | 3 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All participants who were allocated to receive treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-2206 45 mg QOD+Carboplatin+Paclitaxel | MK-2206 60 mg QOD+Carboplatin+Paclitaxel | MK-2206 90 mg Q3W+Carboplatin+Paclitaxel | MK-2206 135 mg Q3W+Carboplatin+Paclitaxel | MK-2206 200 mg Q3W+Carboplatin+Paclitaxel | MK-2206 45 mg QOD+Docetaxel 75 mg/m^2 | MK-2206 90 mg Q3W+Docetaxel 60 mg/m^2 | MK-2206 135 mg Q3W+Docetaxel 60 mg/m^2 | MK-2206 200 mg Q3W+Docetaxel 60 mg/m^2 | MK-2206 45 mg QOD+Erlotinib 100 mg | MK-2206 45 mg QOD+Erlotinib 150 mg | MK-2206 135 mg QW+Erlotinib 100 mg | MK-2206 135 mg QW+Erlotinib 150 mg | Total
Number analyzed (Participants) | 7 | 9 | 6 | 5 | 6 | 5 | 3 | 5 | 4 | 9 | 4 | 6 | 8 | 77
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.6 (15.3) | 58.4 (13.6) | 56.2 (10.4) | 63.6 (7.8) | 38.8 (12.4) | 57.4 (19.7) | 64.7 (12.0) | 57.4 (8.0) | 54.0 (9.4) | 61.6 (6.1) | 61.0 (6.4) | 55.7 (12.7) | 54.1 (10.9) | 56.2 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 2 | 4 | 1 | 2 | 1 | 4 | 3 | 2 | 1 | 2 | 4 | 36
  Male | 3 | 3 | 4 | 1 | 5 | 3 | 2 | 1 | 1 | 7 | 3 | 4 | 4 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  White | 7 | 8 | 6 | 5 | 4 | 4 | 3 | 5 | 4 | 8 | 4 | 6 | 8 | 72
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Dose Limiting Toxicity (DLT) During Cycle 1
Description: A DLT was any of the following deemed drug related by investigator and graded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 criteria: Grade (G)4 hematologic toxicity lasting ≥7 days; G4 thrombocytopenia; G3 or 4 febrile neutropenia and/or infection requiring treatment; G3, 4, 5 non-hematologic toxicity(with the exception of G3 nausea, vomiting, diarrhea, dehydration, or hyperglycemia that as a result of inadequate compliance with supportive care measures; alopecia, inadequately treated hypersensitivity reactions G3 elevated transaminases of ≤1 week in duration); adverse experience (AE) leading to dose reduction; unresolved toxicity causing ≥3 week delay in treatment; ≥G3 hyperglycemia; persistent increases in QTc interval; clinically significant bradycardia; and missing MK-2206 doses due to toxicity. The number of participants who experienced a DLT is presented.
Time Frame: Cycle 1 (Up to 21 days)
Population: All participants that have received one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | MK-2206 45 mg QOD+Carboplatin+Paclitaxel | MK-2206 60 mg QOD+Carboplatin+Paclitaxel | MK-2206 90 mg Q3W+Carboplatin+Paclitaxel | MK-2206 135 mg Q3W+Carboplatin+Paclitaxel | MK-2206 200 mg Q3W+Carboplatin+Paclitaxel | MK-2206 45 mg QOD+Docetaxel 75 mg/m^2 | MK-2206 90 mg Q3W+Docetaxel 60 mg/m^2 | MK-2206 135 mg Q3W+Docetaxel 60 mg/m^2 | MK-2206 200 mg Q3W+Docetaxel 60 mg/m^2 | MK-2206 45 mg QOD+Erlotinib 100 mg | MK-2206 45 mg QOD+Erlotinib 150 mg | MK-2206 135 mg QW+Erlotinib 100 mg | MK-2206 135 mg QW+Erlotinib 150 mg
Number analyzed (Participants) | 6 | 9 | 5 | 5 | 6 | 5 | 3 | 4 | 4 | 9 | 4 | 6 | 6
Participants | 1 | 2 | 1 | 1 | 2 | 3 | 0 | 0 | 1 | 2 | 1 | 0 | 1

2. Primary Outcome: Maximum Tolerated Dose (MTD) of MK-2206 Administered Every Other Day (QOD) in Combination With Carboplatin and Paclitaxel
Description: Participants received MK-2206 (45 or 60 mg) administered PO on Days 1, 3, 5, and 7 in combination with carboplatin AUC 6 and paclitaxel 200 mg/m^2 administered IV on Day 1 of each 21-day cycle. The MTD was determined by the number of participants who experienced a dose limiting toxicity (DLT). DLT was defined using the NCI CTCAE version 3.0 criteria. See primary DLT outcome measure for the DLT definition. The MTD was defined as the dose level, at which the percentage of patients who experienced a DLT rate in Cycle 1 that was closest to 30%. A minimum of 13 participants were required to be enrolled per dose to calculate DLT. If the DLT threshold or enrollment quota per dose were not reached then the MTD could not be determined.
Time Frame: Cycle 1 (Up to 21 days)
Population: All participants who received MK-2206 QOD+carboplatin+paclitaxel and had a DLT in Cycle 1 or received 90% of the planned doses and completed all safety evaluations ≤21 days after the first administration of treatment without experiencing a DLT. MTD could not be determined according to pre-defined protocol criteria based on the enrollment number.
Measure: Number; unit: mg
Groups:
- MK-2206 Administered QOD+Carboplatin+Paclitaxel: Participants received MK-2206 45 mg or 60 mg administered PO on Days 1, 3, 5, and 7 in combination with carboplatin AUC 6 and paclitaxel 200 mg/m^2 administered IV on Day 1 of each 21-day cycle.
Arm/Group | MK-2206 Administered QOD+Carboplatin+Paclitaxel
Number analyzed (Participants) | 9
mg | NA — MTD could not be determined

3. Primary Outcome: MTD of MK-2206 Administered Every Three Weeks (Q3W) in Combination With Carboplatin and Paclitaxel
Description: Participants received MK-2206 (90, 135, or 200 mg) administered PO in combination with carboplatin AUC 6 and paclitaxel 200 mg/m^2 administered IV on Day 1 of each 21-day cycle. The MTD was determined by the number of participants who experienced a DLT. DLT was defined using the NCI CTCAE version 3.0 criteria. See primary DLT outcome measure for the DLT definition. The MTD was defined as the dose level, at which the percentage of patients who experienced a DLT rate in Cycle 1 that was closest to 30%. A minimum of 13 participants were required to be enrolled per dose to calculate DLT. If the DLT threshold or enrollment quota per dose were not reached then the MTD could not be determined.
Time Frame: Cycle 1 (up to 21 days)
Population: All participants who received MK-2206 Q3W+carboplatin+paclitaxel and had a DLT in Cycle 1 or received 90% of the planned doses and completed all safety evaluations ≤21 days after the first administration of treatment without experiencing a DLT. MTD could not be determined according to pre-defined protocol criteria based on the enrollment number.
Measure: Number; unit: mg
Groups:
- MK-2206 Administered Q3W+Carboplatin+Paclitaxel: Participants received MK-2206 90 mg, 135 mg, or 200 mg administered PO in combination with carboplatin AUC 6 and paclitaxel 200 mg/m^2 administered IV on Day 1 of each 21-day cycle.
Arm/Group | MK-2206 Administered Q3W+Carboplatin+Paclitaxel
Number analyzed (Participants) | 15
mg | NA — MTD could not be determined

4. Primary Outcome: MTD of MK-2206 Administered QOD in Combination With Docetaxel
Description: Participants received MK-2206 45 mg administered PO on Days 1, 3, 5, and 7 in combination with Docetaxel 75 mg/m^2 administered IV on Day 1 of each 21-day cycle. Participants also received an oral corticosteroid PO daily. The MTD was determined by the number of participants who experienced a DLT. DLT was defined using the NCI CTCAE version 3.0 criteria. See primary DLT outcome measure for the DLT definition. The MTD was defined as the dose level, at which the percentage of patients who experienced a DLT rate in Cycle 1 that was closest to 30%. A minimum of 13 participants were required to be enrolled per dose to calculate DLT. If the DLT threshold or enrollment quota per dose were not reached then the MTD could not be determined.
Time Frame: Cycle 1 (up to 21 days)
Population: All participants who received MK-2206 QOD+docetaxel and had a DLT in Cycle 1 or received 90% of the planned doses and completed all safety evaluations ≤21 days after the first administration of treatment without experiencing a DLT. MTD could not be determined according to pre-defined protocol criteria based on the enrollment number.
Measure: Number; unit: mg
Groups:
- MK-2206 Administered QOD+Docetaxel: Participants received MK-2206 45 mg administered PO on Days 1, 3, 5, and 7 in combination with Docetaxel 75 mg/m^2 administered IV on Day 1 of each 21-day cycle. Participants also received an oral corticosteroid PO daily.
Arm/Group | MK-2206 Administered QOD+Docetaxel
Number analyzed (Participants) | 5
mg | NA — MTD could not be determined

5. Primary Outcome: MTD of MK-2206 Administered Q3W in Combination With Docetaxel
Description: Participants received MK-2206 (90, 135, or 200 mg) administered PO on Day 1 in combination with Docetaxel 60 mg/m^2 administered IV on Day 1 of each 21-day cycle. Participants also received an oral corticosteroid PO daily. The MTD was determined by the number of participants who experienced a DLT. DLT was defined using the NCI CTCAE version 3.0 criteria. See primary DLT outcome measure for the DLT definition. The MTD was defined as the dose level, at which the percentage of patients who experienced a DLT rate in Cycle 1 that was closest to 30%. A minimum of 13 participants were required to be enrolled per dose to calculate DLT. If the DLT threshold or enrollment quota per dose were not reached then the MTD could not be determined.
Time Frame: Cycle 1 (up to 21 days)
Population: All participants who received MK-2206 Q3W+docetaxel and had a DLT in Cycle 1 or received 90% of the planned doses and completed all safety evaluations ≤21 days after the first administration of treatment without experiencing a DLT. MTD could not be determined according to pre-defined protocol criteria based on the enrollment number.
Measure: Number; unit: mg
Groups:
- MK-2206 Administered Q3W+Docetaxel: Participants received MK-2206 90 mg, 135 mg or 200 mg administered PO on Day 1 in combination with Docetaxel 60 mg/m^2 administered IV on Day 1 of each 21-day cycle. Participants also received an oral corticosteroid PO daily.
Arm/Group | MK-2206 Administered Q3W+Docetaxel
Number analyzed (Participants) | 10
mg | NA — MTD could not be determined

6. Primary Outcome: MTD of MK-2206 Administered QOD in Combination With Erlotinib
Description: Participants received MK-2206 45 mg administered PO every other day (Days 1, 3, 5, 7, 9, 11, 13, 15, 17, 19 and 21) in combination with Erlotinib (100 or 150 mg) administered PO once every day of each 21-day cycle. The MTD was determined by the number of participants who experienced a DLT. DLT was defined using the NCI CTCAE version 3.0 criteria. See primary DLT outcome measure for the DLT definition. The MTD was defined as the dose level, at which the percentage of patients who experienced a DLT rate in Cycle 1 that was closest to 30%. A minimum of 13 participants were required to be enrolled per dose to calculate DLT. If the DLT threshold or enrollment quota per dose were not reached then the MTD could not be determined.
Time Frame: Cycle 1 (up to 21 days)
Population: All participants who received MK-2206 QOD+erlotinib and had a DLT in Cycle 1 or received 90% of the planned doses and completed all safety evaluations ≤21 days after the first administration of treatment without experiencing a DLT. MTD could not be determined according to pre-defined protocol criteria based on the enrollment number.
Measure: Number; unit: mg
Groups:
- MK-2206 Administered QOD+Erlotinib: Participants received MK-2206 45 mg administered PO every other day (Days 1, 3, 5, 7, 9, 11, 13, 15, 17, 19 and 21) in combination with Erlotinib 100 mg or 150 mg administered PO once every day of each 21-day cycle.
Arm/Group | MK-2206 Administered QOD+Erlotinib
Number analyzed (Participants) | 11
mg | NA — MTD could not be determined

7. Primary Outcome: MTD of MK-2206 Administered Once Every Week (QW) in Combination With Erlotinib
Description: Participants received MK-2206 135 mg administered PO on Days 1, 8 and 15 in combination with Erlotinib (100 or 150 mg) administered PO once every day of each 21-day cycle. The MTD was determined by the number of participants who experienced a DLT. DLT was defined using the NCI CTCAE version 3.0 criteria. See primary DLT outcome measure for the DLT definition. The MTD was defined as the dose level, at which the percentage of patients who experienced a DLT rate in Cycle 1 that was closest to 30%. A minimum of 13 participants were required to be enrolled per dose to calculate DLT. If the DLT threshold or enrollment quota per dose were not reached then the MTD could not be determined.
Time Frame: Cycle 1 (up to 21 days)
Population: All participants who received MK-2206 QW+erlotinib and had a DLT in Cycle 1 or received 90% of the planned doses and completed all safety evaluations ≤21 days after the first administration of treatment without experiencing a DLT. MTD could not be determined according to pre-defined protocol criteria based on the enrollment number.
Measure: Number; unit: mg
Groups:
- MK-2206 Administered QW+Erlotinib: Participants received MK-2206 135 mg administered PO on Days 1, 8 and 15 in combination with Erlotinib 100 mg or 150 mg administered PO once every day of each 21-day cycle.
Arm/Group | MK-2206 Administered QW+Erlotinib
Number analyzed (Participants) | 9
mg | NA — MTD could not be determined

8. Primary Outcome: Maximum Plasma Concentration of MK-2206 (Cmax)
Description: Blood samples are to be collected at specified time points according to arm and schedule: QOD schedule for MK-2206+carboplatin+paclitaxel and MK-2206+docetaxel (Cycle 1 Day 1: predose and 2, 4, 6, 10, 24, 48 hours(h) postdose); Q3W schedule MK-2206+carboplatin+paclitaxel and MK-2206+docetaxel (Cycle 1 Day 1: predose and 2, 4, 6, 10, 24, 48, 96h postdose); QOD schedule for the MK-2206+erlotinib (Cycle 1 Day 1: predose and 2, 4, 6, 10, 24, 48h postdose); and QW schedule for MK-2206+erlotinib (Cycles 1 Day 1: predose and 2, 4, 6, 10, 24, 48, 96h postdose) for the determination of MK-2206 Cmax after Dose 1. The Cmax of MK-2206 after Dose 1 will be presented.
Time Frame: At designated time points on Cycle 1 Day 1 (Up to 96 hours)
Population: All participants who received MK-2206 on Cycle 1 Day 1 and had blood samples drawn for the PK parameter being analyzed
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | MK-2206 45 mg QOD+Carboplatin+Paclitaxel | MK-2206 60 mg QOD+Carboplatin+Paclitaxel | MK-2206 90 mg Q3W+Carboplatin+Paclitaxel | MK-2206 135 mg Q3W+Carboplatin+Paclitaxel | MK-2206 200 mg Q3W+Carboplatin+Paclitaxel | MK-2206 45 mg QOD+Docetaxel 75 mg/m^2 | MK-2206 90 mg Q3W+Docetaxel 60 mg/m^2 | MK-2206 135 mg Q3W+Docetaxel 60 mg/m^2 | MK-2206 200 mg Q3W+Docetaxel 60 mg/m^2 | MK-2206 45 mg QOD+Erlotinib 100 mg | MK-2206 45 mg QOD+Erlotinib 150 mg | MK-2206 135 mg QW+Erlotinib 100 mg | MK-2206 135 mg QW+Erlotinib 150 mg
Number analyzed (Participants) | 6 | 8 | 5 | 5 | 6 | 5 | 3 | 3 | 4 | 9 | 4 | 6 | 6
nmol/L | 57.7 (13.8) | 88.3 (24.2) | 144 (57.0) | 247 (52.5) | 431 (249) | 42.9 (13.3) | 106 (42.5) | 278 (35.5) | 287 (67.6) | 48.8 (11.2) | 65.6 (29.3) | 212 (75.9) | 244 (84.2)

9. Primary Outcome: Time to Maximum Plasma Concentration of MK-2206 (Tmax)
Description: Blood samples are to be collected at specified time points according to arm and schedule: QOD schedule for MK-2206+carboplatin+paclitaxel and MK-2206+docetaxel (Cycle 1 Day 1: predose and 2, 4, 6, 10, 24, 48 hours(h) postdose); Q3W schedule MK-2206+carboplatin+paclitaxel and MK-2206+docetaxel (Cycle 1 Day 1: predose and 2, 4, 6, 10, 24, 48, 96h postdose); QOD schedule for the MK-2206+erlotinib (Cycle 1 Day 1: predose and 2, 4, 6, 10, 24, 48h postdose); and QW schedule for MK-2206+erlotinib (Cycles 1 Day 1: predose and 2, 4, 6, 10, 24, 48, 96h postdose) for the determination of MK-2206 Tmax after Dose 1. The Tmax of MK-2206 after Dose 1 will be presented.
Time Frame: At designated time points on Cycle 1 Day 1 (Up to 96 hours)
Population: All participants who received MK-2206 on Cycle 1 Day 1 and had blood samples drawn for the PK parameter being analyzed
Measure: Median (Full Range); unit: hours
Arm/Group | MK-2206 45 mg QOD+Carboplatin+Paclitaxel | MK-2206 60 mg QOD+Carboplatin+Paclitaxel | MK-2206 90 mg Q3W+Carboplatin+Paclitaxel | MK-2206 135 mg Q3W+Carboplatin+Paclitaxel | MK-2206 200 mg Q3W+Carboplatin+Paclitaxel | MK-2206 45 mg QOD+Docetaxel 75 mg/m^2 | MK-2206 90 mg Q3W+Docetaxel 60 mg/m^2 | MK-2206 135 mg Q3W+Docetaxel 60 mg/m^2 | MK-2206 200 mg Q3W+Docetaxel 60 mg/m^2 | MK-2206 45 mg QOD+Erlotinib 100 mg | MK-2206 45 mg QOD+Erlotinib 150 mg | MK-2206 135 mg QW+Erlotinib 100 mg | MK-2206 135 mg QW+Erlotinib 150 mg
Number analyzed (Participants) | 6 | 8 | 5 | 5 | 6 | 5 | 3 | 3 | 4 | 9 | 4 | 6 | 6
hours | 4.0 [4.0 to 6.0] | 8.0 [6.0 to 10.0] | 6.0 [4.0 to 10.0] | 10.0 [6.0 to 10.0] | 5.0 [4.0 to 10.0] | 6.0 [4.0 to 10.0] | 4.0 [4.0 to 10.0] | 6.0 [4.0 to 10.0] | 6.0 [4.0 to 6.0] | 6.0 [4.0 to 10.0] | 7.0 [4.0 to 24.0] | 6.0 [2.0 to 6.0] | 4.0 [4.0 to 10.0]

10. Primary Outcome: Minimum Plasma Concentration of MK-2206 (Ctrough)
Description: Blood samples are to be collected at specified time points according to arm and schedule: QOD schedule for MK-2206+carboplatin+paclitaxel and MK-2206+docetaxel (Cycle 1 Day 1: predose and 2, 4, 6, 10, 24, 48 hours(h) postdose); Q3W schedule MK-2206+carboplatin+paclitaxel and MK-2206+docetaxel (Cycle 1 Day 1: predose and 2, 4, 6, 10, 24, 48h postdose); QOD schedule for the MK-2206+erlotinib (Cycle 1 Day 1: predose and 2, 4, 6, 10, 24, 48h postdose); and QW schedule for MK-2206+erlotinib (Cycles 1 Day 1: predose and 2, 4, 6, 10, 24, 48h postdose) for the determination of MK-2206 Ctrough after Dose 1. The Ctrough after Dose 1 is presented and is the 48-hour postdose concentration.
Time Frame: At designated time points on Cycle 1 Day 1 (Up to 48 hours)
Population: All participants who received MK-2206 on Cycle 1 Day 1 and had blood samples drawn for the PK parameter being analyzed
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | MK-2206 45 mg QOD+Carboplatin+Paclitaxel | MK-2206 60 mg QOD+Carboplatin+Paclitaxel | MK-2206 90 mg Q3W+Carboplatin+Paclitaxel | MK-2206 135 mg Q3W+Carboplatin+Paclitaxel | MK-2206 200 mg Q3W+Carboplatin+Paclitaxel | MK-2206 45 mg QOD+Docetaxel 75 mg/m^2 | MK-2206 90 mg Q3W+Docetaxel 60 mg/m^2 | MK-2206 135 mg Q3W+Docetaxel 60 mg/m^2 | MK-2206 200 mg Q3W+Docetaxel 60 mg/m^2 | MK-2206 45 mg QOD+Erlotinib 100 mg | MK-2206 45 mg QOD+Erlotinib 150 mg | MK-2206 135 mg QW+Erlotinib 100 mg | MK-2206 135 mg QW+Erlotinib 150 mg
Number analyzed (Participants) | 6 | 8 | 5 | 5 | 6 | 5 | 3 | 1 | 4 | 9 | 4 | 6 | 6
nmol/L | 24.9 (10.7) | 40.6 (11.2) | 1.36 (0.898) | 4.67 (3.33) | 2.21 (1.04) | 17.1 (3.66) | 2.27 (1.04) | 3.80 (NA) — Standard deviation could not be calculated for 1 participant | 3.24 (0.638) | 23.8 (8.12) | 36.8 (10.6) | 96.6 (43.6) | 95.5 (43.1)

11. Primary Outcome: Area Under the MK-2206 Concentration Versus Time Curve From Time Zero to 48 Hours Postdose (AUC 0-48h)
Description: Blood samples are to be collected at specified time points according to arm and schedule: QOD schedule for MK-2206+carboplatin+paclitaxel and MK-2206+docetaxel (Cycle 1 Day 1: predose and 2, 4, 6, 10, 24, 48 hours(h) postdose); Q3W schedule MK-2206+carboplatin+paclitaxel and MK-2206+docetaxel (Cycle 1 Day 1: predose and 2, 4, 6, 10, 24, 48h postdose); QOD schedule for the MK-2206+erlotinib (Cycle 1 Day 1: predose and 2, 4, 6, 10, 24, 48h postdose); and QW schedule for MK-2206+erlotinib (Cycles 1 Day 1: predose and 2, 4, 6, 10, 24, 48h postdose) for the determination of MK-2206 AUC0-48h after Dose 1. The AUC0-48h after Dose 1 is presented.
Time Frame: At designated time points on Cycle 1 Day 1 (Up to 48 hours)
Population: All participants who received MK-2206 on Cycle 1 Day 1 and had blood samples drawn for the PK parameter being analyzed
Measure: Mean (Standard Deviation); unit: nmol•hr/L
Arm/Group | MK-2206 45 mg QOD+Carboplatin+Paclitaxel | MK-2206 60 mg QOD+Carboplatin+Paclitaxel | MK-2206 90 mg Q3W+Carboplatin+Paclitaxel | MK-2206 135 mg Q3W+Carboplatin+Paclitaxel | MK-2206 200 mg Q3W+Carboplatin+Paclitaxel | MK-2206 45 mg QOD+Docetaxel 75 mg/m^2 | MK-2206 90 mg Q3W+Docetaxel 60 mg/m^2 | MK-2206 135 mg Q3W+Docetaxel 60 mg/m^2 | MK-2206 200 mg Q3W+Docetaxel 60 mg/m^2 | MK-2206 45 mg QOD+Erlotinib 100 mg | MK-2206 45 mg QOD+Erlotinib 150 mg | MK-2206 135 mg QW+Erlotinib 100 mg | MK-2206 135 mg QW+Erlotinib 150 mg
Number analyzed (Participants) | 6 | 8 | 5 | 5 | 6 | 5 | 3 | 3 | 4 | 9 | 4 | 6 | 6
nmol•hr/L | 1630 (496) | 2700 (619) | 4130 (1520) | 7420 (1250) | 9730 (2320) | 1320 (395) | 3000 (1250) | 8090 (542) | 7690 (1550) | 1460 (417) | 2110 (637) | 6420 (2760) | 6560 (2650)

12. Secondary Outcome: Number of Participants Who Had a Tumor Response of Complete Response (CR) or Partial Response (PR)
Description: Tumor response was assessed using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) and was recorded from the start of the study treatment until the end of treatment. Response categories included: Complete Response (CR): disappearance of all target lesions and Partial Response (PR): at least a 30% decrease in the sum of diameters of target lesions. The number of participants who had a tumor response of either CR or PR is presented.
Time Frame: Up to approximately 4 months (6 cycles)
Population: All participants who received at least one dose of study treatment and had measurable disease at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-2206 45 mg QOD+Carboplatin+Paclitaxel | MK-2206 60 mg QOD+Carboplatin+Paclitaxel | MK-2206 90 mg Q3W+Carboplatin+Paclitaxel | MK-2206 135 mg Q3W+Carboplatin+Paclitaxel | MK-2206 200 mg Q3W+Carboplatin+Paclitaxel | MK-2206 45 mg QOD+Docetaxel 75 mg/m^2 | MK-2206 90 mg Q3W+Docetaxel 60 mg/m^2 | MK-2206 135 mg Q3W+Docetaxel 60 mg/m^2 | MK-2206 200 mg Q3W+Docetaxel 60 mg/m^2 | MK-2206 45 mg QOD+Erlotinib 100 mg | MK-2206 45 mg QOD+Erlotinib 150 mg | MK-2206 135 mg QW+Erlotinib 100 mg | MK-2206 135 mg QW+Erlotinib 150 mg
Number analyzed (Participants) | 6 | 9 | 5 | 5 | 6 | 5 | 3 | 4 | 4 | 9 | 4 | 6 | 6
Participants | 1 | 3 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 14 months (Up to 30 days after last dose of study treatment)
Description: All participants who received at least one dose of study treatment
Groups:
- MK-2206 45 mg QOD+Docetaxel 75 mg/m2: Participants received MK-2206 45 mg administered PO on Days 1, 3, 5, and 7 in combination with Docetaxel 75 mg/m^2 administered IV on Day 1 of each 21-day cycle. Participants also received an oral corticosteroid PO daily.
- MK-2206 90 mg Q3W+Docetaxel 60 mg/m2: Participants received MK-2206 90 mg administered PO on Day 1 in combination with Docetaxel 60 mg/m^2 administered IV on Day 1 of each 21-day cycle. Participants also received an oral corticosteroid PO daily.
- MK-2206 135 mg Q3W+Docetaxel 60 mg/m2: Participants received MK-2206 135 mg administered PO on Day 1 in combination with Docetaxel 60 mg/m^2 administered IV on Day 1 of each 21-day cycle. Participants also received an oral corticosteroid PO daily.
- MK-2206 200 mg Q3W+Docetaxel 60 mg/m2: Participants received MK-2206 200 mg administered PO on Day 1 in combination with Docetaxel 60 mg/m^2 administered IV on Day 1 of each 21-day cycle. Participants also received an oral corticosteroid PO daily.
Arm/Group | MK-2206 45 mg QOD+Carboplatin+Paclitaxel | MK-2206 60 mg QOD+Carboplatin+Paclitaxel | MK-2206 90 mg Q3W+Carboplatin+Paclitaxel | MK-2206 135 mg Q3W+Carboplatin+Paclitaxel | MK-2206 200 mg Q3W+Carboplatin+Paclitaxel | MK-2206 45 mg QOD+Docetaxel 75 mg/m2 | MK-2206 90 mg Q3W+Docetaxel 60 mg/m2 | MK-2206 135 mg Q3W+Docetaxel 60 mg/m2 | MK-2206 200 mg Q3W+Docetaxel 60 mg/m2 | MK-2206 45 mg QOD+Erlotinib 100 mg | MK-2206 45 mg QOD+Erlotinib 150 mg | MK-2206 135 mg QW+Erlotinib 100 mg | MK-2206 135 mg QW+Erlotinib 150 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 1/9 | 0/5 | 0/5 | 0/6 | 1/5 | 0/3 | 0/4 | 0/4 | 1/9 | 0/4 | 1/6 | 1/6
Serious Adverse Events (participants affected / at risk) | 2/6 | 8/9 | 3/5 | 1/5 | 2/6 | 5/5 | 1/3 | 3/4 | 3/4 | 6/9 | 1/4 | 4/6 | 5/6
Other Adverse Events (participants affected / at risk) | 6/6 | 8/9 | 5/5 | 5/5 | 5/6 | 5/5 | 3/3 | 3/4 | 4/4 | 9/9 | 4/4 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-2206 45 mg QOD+Carboplatin+Paclitaxel (N=6) | MK-2206 60 mg QOD+Carboplatin+Paclitaxel (N=9) | MK-2206 90 mg Q3W+Carboplatin+Paclitaxel (N=5) | MK-2206 135 mg Q3W+Carboplatin+Paclitaxel (N=5) | MK-2206 200 mg Q3W+Carboplatin+Paclitaxel (N=6) | MK-2206 45 mg QOD+Docetaxel 75 mg/m2 (N=5) | MK-2206 90 mg Q3W+Docetaxel 60 mg/m2 (N=3) | MK-2206 135 mg Q3W+Docetaxel 60 mg/m2 (N=4) | MK-2206 200 mg Q3W+Docetaxel 60 mg/m2 (N=4) | MK-2206 45 mg QOD+Erlotinib 100 mg (N=9) | MK-2206 45 mg QOD+Erlotinib 150 mg (N=4) | MK-2206 135 mg QW+Erlotinib 100 mg (N=6) | MK-2206 135 mg QW+Erlotinib 150 mg (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal vein occlusion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-2206 45 mg QOD+Carboplatin+Paclitaxel (N=6) | MK-2206 60 mg QOD+Carboplatin+Paclitaxel (N=9) | MK-2206 90 mg Q3W+Carboplatin+Paclitaxel (N=5) | MK-2206 135 mg Q3W+Carboplatin+Paclitaxel (N=5) | MK-2206 200 mg Q3W+Carboplatin+Paclitaxel (N=6) | MK-2206 45 mg QOD+Docetaxel 75 mg/m2 (N=5) | MK-2206 90 mg Q3W+Docetaxel 60 mg/m2 (N=3) | MK-2206 135 mg Q3W+Docetaxel 60 mg/m2 (N=4) | MK-2206 200 mg Q3W+Docetaxel 60 mg/m2 (N=4) | MK-2206 45 mg QOD+Erlotinib 100 mg (N=9) | MK-2206 45 mg QOD+Erlotinib 150 mg (N=4) | MK-2206 135 mg QW+Erlotinib 100 mg (N=6) | MK-2206 135 mg QW+Erlotinib 150 mg (N=6)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 5 (11) | 3 (3) | 3 (3) | 1 (1) | 2 (7) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 6 (23) | 4 (9) | 4 (4) | 1 (1) | 1 (3) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (12) | 1 (1) | 1 (1) | 0 (0) | 2 (7) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 5 (13) | 4 (13) | 3 (3) | 1 (1) | 3 (8) | 2 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 5 (10) | 3 (6) | 2 (2) | 1 (1) | 2 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (3) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 4 (6) | 2 (2) | 1 (1) | 2 (3) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 5 (7) | 3 (5) | 4 (6) | 5 (7)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 6 (6) | 3 (4) | 2 (2) | 4 (6) | 2 (2) | 1 (1) | 1 (1) | 2 (3) | 3 (5) | 4 (4) | 1 (3) | 2 (2)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Post-tussive vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal tenesmus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Steatorrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 2 (3) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 4 (6) | 1 (1) | 4 (11) | 3 (4)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 3 (4) | 1 (1) | 3 (3) | 4 (5) | 3 (4) | 1 (1) | 1 (1) | 1 (2) | 4 (5) | 1 (1) | 1 (1) | 0 (0)
Application site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (5) | 6 (7) | 4 (8) | 5 (5) | 1 (1) | 4 (4) | 3 (4) | 2 (2) | 4 (4) | 5 (5) | 3 (3) | 3 (3) | 4 (5)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (4) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ulcer (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pelvic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ear abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood calcium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prothrombin time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3) | 5 (6) | 2 (3) | 3 (4) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 4 (4) | 2 (2) | 4 (5)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 3 (5) | 1 (1) | 0 (0) | 3 (8) | 2 (2) | 1 (2) | 1 (1) | 3 (5) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 2 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (4) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (4) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Akathisia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multifocal motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 4 (4) | 4 (5) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parkinsonism (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (3) | 1 (1) | 1 (3) | 1 (3) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sensory disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonic convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (2) | 0 (0) | 2 (2)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urogenital fistula (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 2 (3) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 5 (5)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (6) | 6 (7) | 5 (5) | 4 (4) | 2 (2) | 3 (4) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (5) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 3 (6) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (7) | 2 (2)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 4 (6) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 4 (6) | 2 (2) | 0 (0) | 1 (1) | 5 (7) | 3 (5) | 4 (12) | 4 (6)
Rash follicular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0)
Rash morbilliform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angiopathy (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Enrollment in this study was discontinued with Amendment 5.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication guidelines.